CLINICAL TRIAL: NCT03866148
Title: Obstructive Sleep Apnoea and Cardiac Arrhythmias and the Impact of an Implantable Loop Recorder
Brief Title: Obstructive Sleep Apnoea and Cardiac Arrhythmias
Acronym: OSCA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FO409918
Record Dates: First submitted 2019-02-13; First posted 2019-03-07 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea; Cardiovascular Diseases; Arrhythmia; Atrial Fibrillation New Onset
Keywords: Atrial Fibrillation; Obstructive Sleep Apnea; Implantable Loop Recorder; Extended Cardiac Monitoring; Matrix Metalloproteinase-9; Interleukin-6; Tumour Necrosis Factor-Alpha; High sensitivity C-Reactive Protein; High sensitivity Troponin-T; Fibroblast Growth Factor-23; Heart Rate Variability; N-Terminal pro B-type Natriuretic Peptide
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cardiovascular Diseases; Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: 2 groups with the intervention the difference.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ILR (Active Comparator): Participants who will receive the Implantable Loop Recorder (Reveal-LINQ) inserted just after baseline. This is single intervention and lasts for 3 years after which the patient has the option to have it removed.
  Interventions: Device: Reveal LINQ
- No ILR (No Intervention): Participants who will not get the Implantable Loop Recorder (Reveal-LINQ).

INTERVENTIONS:
Device: Reveal LINQ — Insertion of monitoring device called Reveal-LINQ (an implantable loop recorder)
  Arms: ILR

SUMMARY:
This study is a prevelance trial looking at how sleep apnoea affects the heart especially heart rhythms.

Previous research shows that patients suffering from sleep apnoea are much more likely to get heart disease and abnormal heart rhythms (arrhythmias). These defects are sometimes missed by the traditional methods of monitoring i.e. 24-hour Holter monitor and ECGs. This means potentially dangerous arrhythmias may not be detected. Additionally, standard therapy for sleep apnoea does not significantly reduce the risk of heart disease.

This study will recruit 200 participants over a period of 18 months. The research team will observe the heart rhythms of sleep apnoea patients by inserting an implantable loop recorder (ILR) in up to 100 participants. The other 100 patients will simply have standard care. This device will monitor the heart continuously for 3 years allowing us to detect abnormal heart rhythms and treat as necessary.

Demonstrating the incidence of arrhythmia can lead onto a larger study which may change future sleep apnoea management improving their cardiovascular outcomes. Other markers of heart disease such as; blood tests, Magnetocardiography and Echocardiography will be performed on participants to shed more light on the mechanisms which link sleep apnoea and heart disease/arrhythmia.

DETAILED DESCRIPTION:
Sleep apnoea affects up to 1.5 million adults in the United Kingdom (UK). This puts this population at risk of reduced oxygen levels during sleep, poor sleep and increased breathing effort . All of the above put stress on the body and are proven to increase the risk of high blood pressure, heart failure and vascular problems. This can lead to strokes, heart disease and death.

Sleep apnoea patients are at much higher risk of abnormal heart rhythms. Even with continuous positive airways pressure (CPAP) treatment (which is the mainstay in sleep apnoea and does help to reduce arrhythmias) patients are still at higher risk of heart disease and stroke.

An implantable loop recorder (Reveal-LINQ) inserted into sleep apnoea patients will be able to continuously monitor a patient's heart rhythm. This will determine the incidence of arrhythmia in sleep apnoea patients. Any significant abnormalities in either arm of the study will be treated as per National Health Service guidelines and best care. The cost associated with this method of intervention will also be considered.

If there is a high prevalence of arrhythmia a future larger trial, involving much larger numbers and multiple centres, could be conducted to demonstrate reduced risk of stroke or heart attack using this method of arrhythmia detection and management.

Cardiovascular biomarkers, cardiac function, autonomic function and magnetocardiography in these patients could shed light on the mechanisms which cause increased cardiovascular morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe sleep apnoea who require CPAP as standard care (AHI >15)
* Patients between the age of 18 and 75

Exclusion Criteria:

* Patients with a diagnosis of atrial fibrillation (AF), atrial flutter and/or ventricular tachycardia (VT)
* Patients with an ILR already in-situ or an established indication for ILR
* Patients with a palliative diagnosis i.e. life expectancy less than 3 years
* Patients who lack capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-03 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of arrhythmia | 3 years
  Incidence of arrhythmia in sleep apnoea patients as recorded by ILR vs a no ILR group
Autonomic function before and after CPAP | 3 years
  Assess the changes to the heart in sleep apnoea patients before and after CPAP in terms of heart rate variability as measured on 24 hour holter monitors. The raw data is taken from the monitor and then analysed manually. The first data set will be from baseline studies which will be compared to studies done at the 1 year follow-up.

SECONDARY OUTCOMES:
Onset and frequency of atrial fibrillation | 3 years
  Explore the onset and frequency of atrial fibrillation in sleep apnoea patients in order to determine what method of detection is efficient and cost effective.
Rate of Cardiovascular Morbidity | 3 years
  Explore the impact of inserting an ILR in patients with sleep apnoea on cardiovascular morbidity (stroke and myocardial infarction) compared to those without ILR
Rate of Cardiovascular Mortality | 3 years
  Explore the impact of inserting an ILR in patients with sleep apnoea on cardiovascular mortality (stroke and/or myocardial infarction resulting in death) compared to those without ILR
Cardiovascular biomarkers before and after CPAP | 3 years
  Explore the changes to the heart in sleep apnoea patients before and after CPAP in terms of vascular biomarkers - high sensitivity C-Reactive Protein, high sensitivity Troponin-T, N-terminal pro B-type Natriuretic Peptide, Tumour Necrosis Factor-alpha, Matrix Metalloproteinase-9, Interleukin-6, Fibroblast Growth Factor-23. The first data set will be from baseline studies which will be compared to studies done at the 1 year follow-up.
Echocardiography before and after CPAP | 3 years
  Explore the changes to the heart in sleep apnoea patients before and after CPAP in terms of echocardiogram measures.
Quality of life: EQ-5D-5L questionnaire | 3 years
  Quality of life measures before and after CPAP as measured by the EQ-5D 5 level questionnaire. This measures various quality of life points from a scale of 1-5. 1 represents poor quality of life and 5 represents good quality of life for each factor. This data will be analysed as per the EuroQol algorithm. The first data set will be from baseline studies which will be compared to studies done at the 1 year follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Coventry & Warwickshire, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yeung C, Drew D, Hammond S, Hopman WM, Redfearn D, Simpson C, Abdollah H, Baranchuk A. Extended Cardiac Monitoring in Patients With Severe Sleep Apnea and No History of Atrial Fibrillation (The Reveal XT-SA Study). Am J Cardiol. 2018 Dec 1;122(11):1885-1889. doi: 10.1016/j.amjcard.2018.08.032. Epub 2018 Sep 7. PMID 30274768
- [Background] McEvoy RD, Antic NA, Heeley E, Luo Y, Ou Q, Zhang X, Mediano O, Chen R, Drager LF, Liu Z, Chen G, Du B, McArdle N, Mukherjee S, Tripathi M, Billot L, Li Q, Lorenzi-Filho G, Barbe F, Redline S, Wang J, Arima H, Neal B, White DP, Grunstein RR, Zhong N, Anderson CS; SAVE Investigators and Coordinators. CPAP for Prevention of Cardiovascular Events in Obstructive Sleep Apnea. N Engl J Med. 2016 Sep 8;375(10):919-31. doi: 10.1056/NEJMoa1606599. Epub 2016 Aug 28. PMID 27571048
- [Background] Javaheri S, Barbe F, Campos-Rodriguez F, Dempsey JA, Khayat R, Javaheri S, Malhotra A, Martinez-Garcia MA, Mehra R, Pack AI, Polotsky VY, Redline S, Somers VK. Sleep Apnea: Types, Mechanisms, and Clinical Cardiovascular Consequences. J Am Coll Cardiol. 2017 Feb 21;69(7):841-858. doi: 10.1016/j.jacc.2016.11.069. PMID 28209226
- [Derived] He H, Lachlan T, Chandan N, Lim VG, Kimani P, Ng GA, Ali A, Randeva H, Osman F. Obstructive Sleep Apnoea and Cardiac Arrhythmias (OSCA) trial: a nested cohort study using injectable loop recorders and Holter monitoring in patients with obstructive sleep apnoea. BMJ Open. 2023 Feb 15;13(2):e070884. doi: 10.1136/bmjopen-2022-070884. PMID 36792325